CLINICAL TRIAL: NCT03616470
Title: A Phase III Randomized, Double-Blind Trial to Evaluate the Efficacy of Uproleselan Administered With Chemotherapy Versus Chemotherapy Alone in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Study to Determine the Efficacy of Uproleselan (GMI-1271) in Combination With Chemotherapy to Treat Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial failed to meet primary endpoint.
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMI-1271-301
Record Dates: First submitted 2018-07-26; First posted 2018-08-06 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; AML; Relapsed AML; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — uproleselan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Uproleselan (GMI-1271) (Experimental): Uproleselan in combination with mitoxantrone, etoposide and cytarabine (MEC) or fludarabine, cytarabine and idarubicin (FAI)
  Interventions: Drug: Uproleselan
- Placebo (Saline, 0.9% Sodium Chloride) (Placebo Comparator): Placebo in combination with mitoxantrone, etoposide and cytarabine (MEC) or fludarabine, cytarabine and idarubicin (FAI)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Uproleselan — A rationally designed E-selectin antagonist used to inhibit binding of cells to E-selectin
  Arms: Uproleselan (GMI-1271)
Drug: Placebo — Saline, 0.9% Sodium Chloride
  Arms: Placebo (Saline, 0.9% Sodium Chloride)

SUMMARY:
This study will evaluate the efficacy of uproleselan (GMI-1271), a specific E-selectin antagonist, in combination with chemotherapy to treat relapsed/refractory AML, compared to chemotherapy alone. The safety of uproleselan when given with chemotherapy will also be investigated in patients with relapsed/refractory AML

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years and ≤75 years in age
* Patients with relapsed or refractory AML
* No more than one prior stem cell transplant
* Has not received the chemotherapy regimen to be used for induction on this trial
* Is considered medically eligible to receive the chemotherapy regimen to be used for induction on this trial

Exclusion Criteria:

* Patients with acute promyelocytic leukemia, acute leukemia of ambiguous lineage (biphenotypic leukemia), chronic myeloid leukemia with myeloid blast crisis, or secondary refractory AML.
* Active signs or symptoms of CNS involvement by malignancy.
* Stem cell transplantation ≤4 months prior to dosing.
* Any immunotherapy or radiotherapy therapy within 28 days of dosing; any other experimental therapy or chemotherapy within 14 days of dosing.
* Prior use of G-CSF, CM-CSF or plerixafor within 7 days of dosing.
* Inadequate organ function.
* Abnormal liver function.
* Known active infection with hepatitis A, B, or C, or human immunodeficiency virus.
* Moderate kidney dysfunction (glomerular filtration rate <45 mL/min).
* Uncontrolled acute life-threatening bacterial, viral, or fungal infection.
* Clinically significant cardiovascular disease.
* Major surgery within 4 weeks of dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Time from the date of randomization into the study to the date of death.

SECONDARY OUTCOMES:
Rate of severe oral mucositis | up to 60 days
  Incidence of severe oral mucositis experienced in patients after treatment.
Overall response rate | Up to 60 days
  Proportion of subjects who achieve a complete remission [CR] or CR with partial recovery [CRh] of blood counts

OTHER OUTCOMES:
Event-free survival | 5 years
  Time from date of randomization into the study to the date of treatment failure, relapse, or death from any cause; whichever occurs first.
Duration of remission | 5 years
  Time from date of first documented remission to date of relapse or death from any cause, whichever occurs first.
Adverse events | up to 5 months
  Frequency, severity, and relatedness of adverse events.
Pharmacokinetic exposure (amount of uproleselan in the blood) | up to 6 days
  The amount of uproleselan in the blood over time.
Event-free survival | 1 year
  Landmark analysis: Time from date of randomization into the study to the date of relapse or death from any cause; whichever occurs first.
Overall survival | 2 years
  Landmark analysis: Time from the date of randomization into the study to the date of death.
Overall survival | 3 years
  Landmark analysis: Time from the date of randomization into the study to the date of death.
Overall survival | 4 years
  Landmark analysis: Time from the date of randomization into the study to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J DeAngelo, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (70):
- United States (30):
  - UC San Diego Moore Cancer Center, La Jolla, California
  - University of California, Los Angeles - UCLA, Los Angeles, California
  - University of California Irvine, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital - Medical Tower, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hudson Valley Cancer Center, Hawthorne, New York
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Health System (DUHS), Durham, North Carolina
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center and James Cancer Hospital, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Vanderbilt-Ingram Cancer Center Clinical Trials Office, Nashville, Tennessee
  - Charles A. Sammons Cancer Center at Dallas, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (6):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Sir Charles Gairdner Hospital, Nedlands, Perth
  - Townsville Hospital, Douglas, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Cancer Clinical Trials Centre (CCTC), Heidelberg, Victoria
- Canada (6):
  - Tom Baker Cancer Center, Calgary, Alberta
  - University of Alberta Princess Margaret Hospital, Edmonton, Alberta
  - The Leukemia/BMT Program of BC Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - University Health Network (UHN) - Princess Margaret Cancer Centre, Toronto, Ontario
- France (7):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche
  - Unité d'Evaluation Thérapeutique en Onco-Hématologie (ETHO), Marseille
  - Saint-Louis Hospital, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
- Galway University Hospital, Galway, Ireland
- Italy (7):
  - IRCCS Casa Sollievo della Sofferenza Hospital, San Giovanni Rotondo, FG
  - Institute of Hematology and Medical Oncology "L. and A. Seràgnoli", Bologna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola
  - Hospital of Ravenna, Ravenna
  - Fondazione Policlinico Tor Vergata, U.O.C. Ematologia, Roma
  - Università Cattolica del Sacro Cuore (UNICATT), Rome
  - Ca' Foncello Hospital, Treviso
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - University Medical Centre Utrecht, Utrecht
- Spain (8):
  - Hospital San Pedro De Alcantra, Cáceres
  - Hospital MDACC, Madrid
  - Hospital Universitario Fundación Jiménez Diaz, Madrid
  - Hospital Virgen de la Victoria, Málaga, Málaga
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - University Hospital of Hospital Marqués de Valdecilla, Santander
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (2):
  - Radcliffe Hospitals and University of Oxford, Oxford, England
  - Cardiff University School of Medicine, Cardiff